CLINICAL TRIAL: NCT06157112
Title: Students' Lifestyle Behaviour and Later Health Care Utilization Due to Musculoskeletal Pain
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Responsible Party: Principal Investigator, Britt Elin Øiestad, Professor, Oslo Metropolitan University
Other Study IDs: 251771
Record Dates: First submitted 2023-11-27; First posted 2023-12-05 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2023-11

CONDITIONS: Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Norwegian University students: Norwegian fulltime University students
  Interventions: Other: Lifestyle behaviour (exposure in a observational study)

INTERVENTIONS:
Other: Lifestyle behaviour (exposure in a observational study) — Lifestyle behaviour, including physical activity, sleep duration, alcohol consumption, smoking, cannabis and other illegal drugs

SUMMARY:
This study aims to assess whether there is an association between students' lifestyle behaviour, in terms of physical activity level, sleep duration, smoking status, alcohol consumption and use of cannabis and other illegal drugs, and later health care utilisation due to musculoskeletal pain. The study will combine data from a national survey in Norway (SHOT2018), in which all full-time university students in Norway were invited, with data from a register on health care utilisation in primary health care.

DETAILED DESCRIPTION:
This study aims to determine:

i) whether male and female university students' lifestyle behaviours, in terms of physical activity level, sleep durance, alcohol consumption, smoking and illicit drug use, are associated with future health care utilisation for musculoskeletal pain, back pain or neck pain, and ii) whether the number of adverse lifestyle behaviours is associated with future health care utilisation for musculoskeletal pain, back pain or neck pain.

Study design and setting:

Cohort study, in which data from the Students' Health and Wellbeing study (SHoT) is merged with data from the Norwegian Register of Primary Health Care (NRPHC).

The eligibility criteria:

Inclusion criteria • Participants of the SHoT2018 study (18-35 years of age)

Exclusion criteria

* Participants studying abroad
* Participants above 35 years of age
* Recent health care utilisation for a musculoskeletal pain diagnosis (the last 12 months prior to the exposure assessment)

Primary outcome:

- Health care utilisation for musculoskeletal pain in primary health care, registered in the NRPHC (follow-up period: 3 years after baseline)

Secondary outcome:

* Health care utilisation for back pain, registered in NRPHC (follow-up period: 3 years after baseline)
* Health care utilisation for neck pain, registered in NRPHC (follow-up period: 3 years after baseline)

Exposures:

* Physical activity, obtained from the SHOT-questionnaire, categorised in accordance with recommendations for weekly physical activity
* Sleep duration, obtained from the SHOT-questionnaire, categorised in accordance with recommendations
* Smoking (yes / no)
* Alcohol consumption (assessed with AUDIT)
* Illegal drug use (categorised in use the last year yes/no)
* Number of adverse lifestyle behaviours (0-5) (low physical activity, short sleep duration, smoking, risky alcohol use, illegal drug use the last year)

Potential confounders:

The following variables will be considered as potential confounders in the analyses: age, financial difficulties, physical health complaints, symptoms of depression and anxiety, BMI, other lifestyle behaviours, consultation frequency irrespective of cause, the last year prior baseline (the last will be used as an indicator of health care seeking behaviour)

Statistical analyses:

3-year incidence rates of health utilisation for musculoskeletal pain, back pain and neck pain will be computed

Crude and adjusted associations between each of the lifestyle behaviours and health care utilisation for musculoskeletal pain, back pain and neck pain will be assessed separately. Also, the association between the number of adverse lifestyle behaviours and musculoskeletal pain, back and neck pain will be assessed in crude and adjusted analyses. Modified Poisson regression will be used to analyse the associations with binary outcomes (health care utilisation for musculoskeletal pain yes/no). To asses the associations with an outcome variable reflecting the number of health care visits for musculoskeletal pain, the exact statistical analysis method will be chosen after inspection of the distribution of the outcome data. All analyses will be conducted stratified by sex.

The following sensitivity analyses will be considered:

* analyses stratified by baseline musculoskeletal pain status
* only including outcome data before 12 March 2020 to assess the associations prior to the Covid 19 restrictions
* excluding participants above 30 years of age to assess the associations in a sample of students withing the "emerging adult" definition (up to 30 years of age)

All analyses will be conducted with STATA statistical software system, version 16 (StataCorp., 2019)

ELIGIBILITY:
Inclusion Criteria:

* All full-time Norwegian University students aged 18 to 35 years of age

Exclusion Criteria:

* students studying abroad
* students above 35 years of age
* students with health care utilisation due to musculoskeletal pain the last 12 months before baseline

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: University full-time students, 18-35 years of age
Sampling Method: Probability Sample
Enrollment: 50054 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2021-04-05 (Actual); Study Completion 2021-04-05 (Actual)

PRIMARY OUTCOMES:
Health care utilisation due to musculoskeletal pain | 3 years (6 Apr 2018 - 6 Apr 2021)
  Visiting a primary health care provider (GP, physiotherapist or chiropractor) due to a musculoskeletal pain diagnosis (yes/no and number of visits)

SECONDARY OUTCOMES:
Health care utilisation due to back pain | 3 years (6 Apr 2018 - 6 Apr 2021)
  Visiting a primary health care provider (GP, physiotherapist or chiropractor) due to a back pain diagnosis
Health care utilisation due to neck pain | 3 years (6 Apr 2018 - 6 Apr 2018)
  Visiting a primary health care provider (GP, physiotherapist or chiropractor) due to a neck pain diagnosis

CONTACTS AND LOCATIONS:
Overall Officials: Britt Elin Øiestad, PhD, Principal Investigator — Oslo Metropolitan University
Locations (1):
- Oslo Metropolitan University, Oslo, Norway, Norway

IPD SHARING:
Plan to Share IPD: No